CLINICAL TRIAL: NCT00348244
Title: A Masked Comparison of Acular LS Plus Steroid Versus Steroid Alone for the Prevention of Macular Leakage in Cataract Patients
Brief Title: Ketorolac vs. Steroid in the Prevention of CME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 5152
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2007-01-17 (Estimated); Status verified 2007-01

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Ketorolac; prednisolone acetate

INTERVENTIONS:
Drug: Ketorolac, Prednisolone Acetate

SUMMARY:
Evaluate if the incidence of sub clinical CME can be significantly reduced by use of peri-operative Acular LS plus Pred Forte when compared with Pred Forte alone in normal cataract patients.

ELIGIBILITY:
Inclusion Criteria:

* · Male or female > 18 years of age scheduled to undergo cataract surgery with surgeon expectation of 20/20 BCVA postoperatively

  * Must be in good general health. Patients with systemic diseases will be enrolled only if there are no ocular manifestations of their disease (ie diabetics with normal retinal exams)
  * Ability to provide informed consent and likely to complete all study visits

Exclusion Criteria:

* · Known contraindication to any study medication or any of their components

  * Uncontrolled systemic disease
  * Required use of ocular medications other than the study medications during the study
  * Abnormal pre-operative OCTs if obtainable
  * Diabetic patients with a history of macular edema or diabetic retinopathy
  * AMD patients with less than a 20/20 surgical outcome expectation, epi-retinal membranes, retinal vein occlusion, or any pre-existing macular disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: John Wittpenn, MD, Principal Investigator — Ophthalmic Consultants of Long Island
Locations (1):
- Dr. Wittpenn, Stony Brook, New York, United States

REFERENCES:
- [Derived] Wittpenn JR, Silverstein S, Heier J, Kenyon KR, Hunkeler JD, Earl M; Acular LS for Cystoid Macular Edema (ACME) Study Group. A randomized, masked comparison of topical ketorolac 0.4% plus steroid vs steroid alone in low-risk cataract surgery patients. Am J Ophthalmol. 2008 Oct;146(4):554-560. doi: 10.1016/j.ajo.2008.04.036. Epub 2008 Jul 2. PMID 18599019